CLINICAL TRIAL: NCT02984267
Title: Use of Ultrasound Guidance to Assist With Labor Epidural Placement in Patients With a BMI ≥40
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas J. Vernon (Other)
Collaborators: West Penn Allegheny Health System (Other)
Responsible Party: Sponsor-Investigator, Thomas J. Vernon, OB Anesthesia Fellow, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OBUS1123
Record Dates: First submitted 2016-11-23; First posted 2016-12-06 (Estimated); Results first posted 2018-07-11 (Actual); Last update posted 2018-07-11 (Actual); Status verified 2018-06

CONDITIONS: Labor Pain
MeSH Terms: conditions — Labor Pain | interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ultrasound Group (Experimental): The interventional group that will have their spine evaluated by ultrasound prior to epidural placement
  Interventions: Device: Ultrasound
- Palpation Group (Other): The control group that will have their epidural placed in the usual fashion based on palpation
  Interventions: Other: Palpation

INTERVENTIONS:
Device: Ultrasound — Using ultrasound guidance to evaluate the spine prior to epidural placement
  Arms: Ultrasound Group
Other: Palpation — Using palpation only to evaluate the spine prior to epidural placement
  Arms: Palpation Group

SUMMARY:
Placement of labor epidurals is a very common daily practice in obstetrical anesthesia. Currently, these epidurals are placed based upon palpation of landmarks to determine midline and the correct spinal level for placement. Palpation of these landmarks can be difficult, however, particularly in morbidly obese patients who have significant amounts of soft tissue overlying them. This study seeks to use ultrasound guidance to examine the spine prior to epidural placement, and see what effects this has compared to palpation alone with respect to procedure time, number of attempts, success rate in the first attempt, failure rate, complication rate, patient anxiety levels, and patient satisfaction levels.

ELIGIBILITY:
Inclusion Criteria:

* Current (pregnant) BMI ≥ 40
* Age ≥ 18
* ASA score of 3 or less
* Full term pregnancy (37 weeks gestational age or greater)

Exclusion Criteria:

* Known scoliosis
* Known contraindications to neuraxial blockade
* Intrauterine fetal demise or non-viable fetus.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-12; Primary Completion 2017-04-15 (Actual); Study Completion 2017-04-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Magee Women's Hospital, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ultrasound Group | Palpation Group
Started | 8 | 10
Completed | 7 | 9
Not Completed | 1 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Ultrasound 43.75% (7/16); Palpation 56.25% (9/16)
Groups:
- Total: Total of all reporting groups
Arm/Group | Ultrasound Group | Palpation Group | Total
Number analyzed (Participants) | 7 | 9 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.3 (4.7) | 29.9 (5.5) | 27.9 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 16
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 6 | 8 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Gravidity [Median (Inter-Quartile Range); unit: Number of pregnancies] | 1 [1 to 2] | 2 [1 to 3] | 2 [1 to 3]
Parity [Median (Inter-Quartile Range); unit: Number of children born] | 0 [0 to 1] | 0 [0 to 1] | 0 [0 to 1]
Estimated gestational age [Mean (Standard Deviation); unit: Weeks] | 39.6 (0.8) | 38.1 (1.1) | 38.7 (1.1)
Weight [Mean (Standard Deviation); unit: kg] | 122.0 (17.1) | 120.6 (15.8) | 121.2 (15.8)
Height [Mean (Standard Deviation); unit: cm] | 163.7 (5.3) | 162.1 (5.3) | 162.8 (5.2)
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 45.6 (7.4) | 45.9 (6.3) | 45.8 (6.6)
American Society of Anesthesiologists (ASA) physical status [Count of Participants; unit: Participants] — ASA1, ASA2, and ASA3 are all categories that participants could fall into based on the status of their overall health. ASA1 indicates a normal, healthy patient. ASA2 indicates a patient with mild systemic disease (examples include but are not limited to pregnancy, current smoker, obesity with a BMI >30 but <40, and well controlled diabetes or hypertension). ASA3 indicates a patient with severe systemic disease (examples include but are not limited to poorly controlled diabetes or hypertension, chronic obstructive pulmonary disorder, morbid obesity with a BMI greater than or equal to 40).
  Participants
    ASA1 | 0 | 0 | 0
    ASA2 | 0 | 0 | 0
    ASA3 | 7 | 9 | 16
External landmarks visible [Count of Participants; unit: Participants] — The back of the patient is visually examined to determine if the outline of the spinous processes of the vertebrae can be seen through the skin.
  Participants
    Yes | 0 | 0 | 0
    No | 7 | 9 | 16
Palpable interspace [Count of Participants; unit: Participants] — A patient has "palpable interspaces" when the spinous processes of the vertebrae, and thus the interspaces between them, can easily be physically felt by the provider through the patient's skin. Population: Palpation was not performed in ultrasound group because only the ultrasound was used to asses location for epidural catheter placement in that group. The number of participants in the ultrasound group reflects only the number analyzed (i.e. 0) and the total number of participants analyzed reflects the total number analyzed (i.e. 9 participants).
  Participants
    number analyzed (Participants) | 0 | 9 | 9
    Yes | 0 | 5 | 5
    No | 0 | 4 | 4

OUTCOME MEASURES:

1. Primary Outcome: Total Time Required for Epidural Catheter Placement
Description: Includes the time required to evaluate the spine (via ultrasound or palpation) plus the time required to successfully place the epidural catheter
Time Frame: Assessed immediately during epidural catheter placement
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Ultrasound Group | Palpation Group
Number analyzed (Participants) | 7 | 9
Minutes | 6.1 (3.5) | 11.0 (5.3)

2. Secondary Outcome: Epidural Procedure Time
Description: Time required to successfully place the epidural catheter
Time Frame: Assessed immediately during epidural catheter placement
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Ultrasound Group | Palpation Group
Number analyzed (Participants) | 7 | 9
Minutes | 4.33 (3.5) | 10.1 (5.4)

3. Secondary Outcome: Number of Attempts at Epidural Catheter Placement
Time Frame: Assessed immediately during epidural catheter placement
Measure: Median (Inter-Quartile Range); unit: Number of attempts
Arm/Group | Ultrasound Group | Palpation Group
Number analyzed (Participants) | 7 | 9
Number of attempts | 1 [1 to 1] | 5 [3 to 5]

4. Secondary Outcome: Number of Participants Who Had Successful Placement of the Epidural Catheter in the First Attempt
Time Frame: Assessed immediately during epidural catheter placement
Measure: Count of Participants; unit: Participants
Arm/Group | Ultrasound Group | Palpation Group
Number analyzed (Participants) | 7 | 9
Participants | 5 | 2

5. Secondary Outcome: Complications
Description: Any epidural related complication noted to occur including a failed epidural, inadvertent dural puncture, or paresthesia will be documented and reported.
Time Frame: Assessed immediately during epidural catheter placement and within 24 hours after delivery
Measure: Number; unit: Complications
Arm/Group | Ultrasound Group | Palpation Group
Number analyzed (Participants) | 7 | 9
Complications | 0 | 4

6. Secondary Outcome: Epidural Failure Rate
Description: Any epidural catheter that fails to provide appropriate analgesia requiring them to be replaced with a new epidural catheter will be documented and reported
Time Frame: Assessed within 24 hours after delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Ultrasound Group | Palpation Group
Number analyzed (Participants) | 7 | 9
Participants | 0 | 0

7. Secondary Outcome: Epidural Catheter Placement Satisfaction Level
Description: Immediately following epidural catheter placement, patients will be asked to rate their satisfaction level during the procedure on a 0-10 scale, with 0 being not at all satisfied, and 10 being extremely satisfied.
Time Frame: Assessed immediately following epidural catheter placement
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Ultrasound Group | Palpation Group
Number analyzed (Participants) | 7 | 9
Units on a scale | 9 (1.2) | 7.3 (2.8)

8. Secondary Outcome: Patient Anxiety Level
Description: Immediately following epidural catheter placement, patients will be asked to rate their anxiety level during the procedure on a 0-10 scale, where 0 is no anxiety at all, and 10 is the worst anxiety imaginable.
Time Frame: Assessed immediately following epidural catheter placement
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Ultrasound Group | Palpation Group
Number analyzed (Participants) | 7 | 9
Units on a scale | 5.4 (1.9) | 6.0 (2.6)

9. Secondary Outcome: Palpation or Ultrasound Time
Description: The time taken to evaluate the spine, either by palpation or ultrasound guidance, and mark the location for epidural catheter insertion
Time Frame: Assessed immediately prior to epidural catheter placement
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Ultrasound Group | Palpation Group
Number analyzed (Participants) | 7 | 9
Minutes | 1.8 (0.6) | 0.9 (0.1)

10. Secondary Outcome: Overall Anesthesia Experience Satisfaction
Description: Within 24 hours after delivery, patients will be given a 13 question survey. The survey is a modified Woman's Views of Birth Labor Satisfaction Questionnaire (WOMBLSQ) which asks patients to rate 13 various satisfaction related statements on a 1-7 scale, with 1 being totally disagree, 4 being neither agree nor disagree, and 7 being totally agree. Each of the 13 questions asked are designed to assess their overall satisfaction with their epidural catheter placement and overall anesthesia care. The total score is reported combining all 13 questions for a possible score range of 13-91. A higher total score indicates a higher overall anesthesia experience satisfaction level. No subscales were used.
Time Frame: Measured within 24 hours of delivery
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Ultrasound Group | Palpation Group
Number analyzed (Participants) | 7 | 9
Units on a scale | 79.1 (11.8) | 74.3 (9.4)

ADVERSE EVENTS:
Time Frame: During the patients current hospitalization (typically 2-3 days)
Description: All study participants were evaluated during and immediately following their epidural catheter procedure, and also later followed up on in person by study personnel within 24 hours of their delivery to assess for any adverse events
Arm/Group | Ultrasound Group | Palpation Group
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/9
Other Adverse Events (participants affected / at risk) | 0/7 | 3/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ultrasound Group (N=7) | Palpation Group (N=9)
Inadvertent dural puncture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Number of participants sustaining an inadvertent dural puncture during the procedure resulting in the formation of a post-dural puncture headache
Paresthesia (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) — Number of patients experiencing a transient paresthesia in their back or leg(s) during epidural catheter placement

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2016-10-01): https://cdn.clinicaltrials.gov/large-docs/67/NCT02984267/SAP_000.pdf
  • Study Protocol (2016-10-01): https://cdn.clinicaltrials.gov/large-docs/67/NCT02984267/Prot_001.pdf